CLINICAL TRIAL: NCT07124520
Title: Normative Ranges of Lingual Strength and Endurance and the Impact of the IOPI Lingual Strength Trainer on Quantitative Functional Outcomes and Patient-Reported Outcomes After Partial Glossectomy or Hemiglossectomy for Oral Tongue Cancer, A Pilot Study
Brief Title: A Study of Tongue Strength and Endurance Using the Iowa Oral Performance Instrument (IOPI) Tongue Strength Trainer in People With Oral Tongue Cance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-162
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Tongue Cancer
Keywords: Tongue Cancer; Oral Tongue Cancer; IOPI Lingual Strength Trainer; Iowa Oral Performance Instrument; Iowa Oral Performance Instrument Tongue Strength Trainer; Memorial Sloan Kettering Cancer Center; 25-162
MeSH Terms: conditions — Tongue Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment Group (Experimental): Standard of care plus intervention with the Iowa Oral Performance Instrument /IOPI. Randomization will be stratified by partial glossectomy versus hemiglossectomy.
  Interventions: Device: Iowa Oral Performance Instrument (IOPI)
- Control Group (No Intervention): Participants will receive standard of care. Randomization will be stratified by partial glossectomy versus hemiglossectomy.

INTERVENTIONS:
Device: Iowa Oral Performance Instrument (IOPI) — The Iowa Oral Performance Instrument/IOPI is an instrument that objectively measures tongue strength using a standard-sized air-filled bulb. An individual presses the bulb against the roof of the mouth with the tongue to generate a pressure measurement in kilopascals (kPa). Maximum tongue strength can be determined using a measure of pressure.
  Arms: Treatment Group

SUMMARY:
The purpose of this study is to learn more about tongue strength and endurance by using the Iowa Oral Performance Instrument (IOPI). The IOPI is a device that measures tongue pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Scheduled to undergo primary surgery for oral tongue cancer (glossectomy types 1 to 3) using any type of closure or reconstruction

Exclusion Criteria:

* Previous radiation therapy to the oral cavity or head and neck
* Previous surgery for oral cavity cancer
* Recurrent oral cavity cancer
* Surgical requirement of extension to involve bone (mandible resection)
* Subtotal or total glossectomy
* Feeding tube dependance prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2028-08-07 (Estimated); Study Completion 2028-08-07 (Estimated)

PRIMARY OUTCOMES:
Tongue strength as measured by Iowa Oral Performance Instrument/IOPI | Up to 6 months
  Define normative ranges in tongue strength using the Iowa Oral Performance Instrument/IOPI in patients with oral tongue cancers undergoing primary surgical resection.
Endurance as measured by Iowa Oral Performance Instrument/IOPI | Up to 6 months
  Define normative ranges in tongue endurance using the Iowa Oral Performance Instrument/IOPI in patients with oral tongue cancers undergoing primary surgical resection.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Cunningham, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memoral Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Consent only), Commack, New York
  - Memoral Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activites), New York, New York
  - Memorial Sloan Kettering Cancer Center @ Nassau (Consent only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org